CLINICAL TRIAL: NCT04703751
Title: Evaluation of the CIRCULATE Catheter for Transcoronary Administration of Pharmacologic and Cell-based Agents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: John Paul II Hospital, Krakow (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIRCULATE catheter evaluation
Record Dates: First submitted 2020-12-31; First posted 2021-01-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Intervention Model Description: Clinical evaluation of the CIRCULATE catheter will be performed in a group of 10 patients. Each will receive intracoronary NTG followed by labelled CardioCell.
  This is a non-randomized study without any requirement for sample size calculation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CIRCULATE Catheter (Experimental): CIRCULATE Catheter will be used to deliver nitroglycerin and CardioCell to evaluate safety and efficacy of the device
  Interventions: Device: Transcoronary delivery of a pharmacological agent (nitroglycerin) and cell based agent (Cardiocell) using the CIRCULATE Catheter

INTERVENTIONS:
Device: Transcoronary delivery of a pharmacological agent (nitroglycerin) and cell based agent (Cardiocell) using the CIRCULATE Catheter — Investigated device - the CIRCULATE Catheter will be introduced, using a standard radial or femoral access and a typical guiding catheter and typical coronary wire, first into the right coronary artery. After that the one dose of NTG (200µg) will be administered followed by a typical angiographic recording to visualize the vasodilatatory effect of the medication. Then CardioCell in doses of 10mln cells each (6.7mL) will be administered transcoronary to each of the coronary arteries (right coronary artery (RCA), LAD, left circumflex (Cx)). Angiography will be performed routinely before and after each product administration.

SUMMARY:
Clinical evaluation of the CIRCULATE catheter involves intracoronary administration of a typical medical agent (nitroglycerin) and a shown-to-be-safe cell-based agent (CardioCell) in patients with a diagnosis of dilated cardiomyopathy (DCM).

DETAILED DESCRIPTION:
The use of adult stem cells from several sources has been shown to improve cardiac function in acute and chronic cardiac disease. Several sources of adult stem cells have been identified including bone marrow, skeletal muscle, blood and adipose tissue. A number of pilot trials using intramyocardial injection of stem cells have shown promising results in patients with chronic myocardial disease in patients with ischemic heart failure , and in patients after an acute myocardial infarction .

The vast majority of research on cell therapies in the treatment of heart diseases focuses mainly on determining the optimal source of cells, their characteristics, and the number of cells in the administered preparation. From a clinical perspective, the method of cell administration is also an important topic.

There are several ways of cell administration that can be used in cell therapy for heart muscle disease. In addition to the intramuscular administration systems, such preparations can be administered directly into the circulation in a more or less selective manner. As no dedicated devices were developed, various types of catheters and microcatheters have been used for transcoronary administration. During the procedure of administering cell preparations by means of a catheter directly to the selected coronary vessel, the flow parameters should be adjusted to minimize the risk of damage to the administered cells.

The CIRCULATE catheter tested in the experiment was designed to increase the efficacy and safety of the cells delivery. It has a reservoir and holes created through which - as shown in preclinical studies - the cells can be delivered without a risk of their damage during delivery.

In addition to the administration of cell therapy, the course of the study is planned to administer the drug - nitroglycerin - one of the most commonly used drugs for coronary administration, recommended during standard angiography of the coronary arteries due to its ability to expand the arterial bed, thus enabling accurate imaging and sizing of the examined arteries.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DCM
* Left ventricular ejection fraction (LVEF) ≤ 45% by echocardiography
* Signed informed consent

Exclusion Criteria:

* Less than 3 months from any substantial cardiac therapeutic intervention (such as, e.g. CRT/ICD fitting)
* Less than 3 months from acute coronary syndrome
* BMI lower than 18 or greater than 45kg/m2
* Severe valvular heart disease or left ventricle aneurysm requiring aneurysmectomy or other structural interventions
* Present candidate for heart transplantation
* Active or any history of malignancy or tumor
* Moderate or severe immunodeficiency
* Chronic immunosuppressive therapy
* Acute or chronic infection
* Coagulopathies
* Known alcohol or drug dependence
* Severe renal dysfunction (eGFR<20mL/min)
* Soft tissue disease or local infection in a place of required artery puncture
* Pregnancy or breastfeeding
* Females of childbearing potential who do not use a highly effective method of contraception, and in absence of a negative highly sensitive urine or serum pregnancy test
* Participation in any other clinical research study that has not reached its primary efficacy endpoint or otherwise would interfere with the patient's participation in this project
* Life expectancy <12 months
* Any concurrent disease or condition that, in the opinion of the investigator, would make the patient unsuitable for participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Device success | During procedure
  Device success, defined as the device introduction, administration of nitroglycerine and cell-based agent, and device removal without complications

SECONDARY OUTCOMES:
Standardized uptake values (SUVs) of 99mTc-HMPAO radiolabelled CardioCell | 1 hour after application
  CardioCell myocardial uptake on a whole-body scan: 50% of cells will be radiolabelled. Standardized uptake values (SUVs) of 99mTc-HMPAO radiolabelled CardioCell in cardiac VOI on a whole-body scan measured using the commercial calculation methods corrected for physical decay and attenuation
Freedom from major adverse cardiovascular events | 24 hours or until hospital discharge, whichever time point is first
  Freedom from periprocedural (during the procedure and 60 minutes thereafter) major adverse cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Musialek, MD, DPhil, Principal Investigator — The John Paul II Hospital
Locations (1):
- Department of Cardiac and Vascular Diseases, John Paul II Hospital, Krakow, Maloplska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Musialek P, Mazurek A, Jarocha D, Tekieli L, Szot W, Kostkiewicz M, Banys RP, Urbanczyk M, Kadzielski A, Trystula M, Kijowski J, Zmudka K, Podolec P, Majka M. Myocardial regeneration strategy using Wharton's jelly mesenchymal stem cells as an off-the-shelf 'unlimited' therapeutic agent: results from the Acute Myocardial Infarction First-in-Man Study. Postepy Kardiol Interwencyjnej. 2015;11(2):100-7. doi: 10.5114/pwki.2015.52282. Epub 2015 Jun 22. PMID 26161101
- [Background] Musialek P, Tracz W, Skotnicki AB, Zmudka K, Pieniazek P, Walter Z, Szostek M, Majka M, Weglarska D, Zalewski J, Olszowska M, Kostkiewicz M, Pasowicz M, Klimeczek P, Przewlocki T. Transcoronary stem cell delivery using physiological endothelium-targeting perfusion technique: the rationale and a pilot study involving a comparison with conventional over-the-wire balloon coronary occlusions in patients after recent myocardial infarction. Kardiol Pol. 2006 May;64(5):489-98; discussion 499. English, Polish. PMID 16752333
- [Background] Musialek P, Tekieli L, Kostkiewicz M, Miszalski-Jamka T, Klimeczek P, Mazur W, Szot W, Majka M, Banys RP, Jarocha D, Walter Z, Krupinski M, Pieniazek P, Olszowska M, Zmudka K, Pasowicz M, Kereiakes DJ, Tracz W, Podolec P, Wojakowski W. Infarct size determines myocardial uptake of CD34+ cells in the peri-infarct zone: results from a study of (99m)Tc-extametazime-labeled cell visualization integrated with cardiac magnetic resonance infarct imaging. Circ Cardiovasc Imaging. 2013 Mar 1;6(2):320-8. doi: 10.1161/CIRCIMAGING.112.979633. Epub 2012 Dec 27. PMID 23271789
- [Background] Musialek P, Tekieli L, Kostkiewicz M, Majka M, Szot W, Walter Z, Zebzda A, Pieniazek P, Kadzielski A, Banys RP, Olszowska M, Pasowicz M, Zmudka K, Tracz W. Randomized transcoronary delivery of CD34(+) cells with perfusion versus stop-flow method in patients with recent myocardial infarction: Early cardiac retention of (9)(9)(m)Tc-labeled cells activity. J Nucl Cardiol. 2011 Feb;18(1):104-16. doi: 10.1007/s12350-010-9326-z. Epub 2010 Dec 14. PMID 21161463
- [Background] Botti C, Negri DR, Seregni E, Ramakrishna V, Arienti F, Maffioli L, Lombardo C, Bogni A, Pascali C, Crippa F, Massaron S, Remonti F, Nerini-Molteni S, Canevari S, Bombardieri E. Comparison of three different methods for radiolabelling human activated T lymphocytes. Eur J Nucl Med. 1997 May;24(5):497-504. doi: 10.1007/BF01267680. PMID 9142729
- [Background] Beeres SL, Bengel FM, Bartunek J, Atsma DE, Hill JM, Vanderheyden M, Penicka M, Schalij MJ, Wijns W, Bax JJ. Role of imaging in cardiac stem cell therapy. J Am Coll Cardiol. 2007 Mar 20;49(11):1137-48. doi: 10.1016/j.jacc.2006.10.072. Epub 2007 Mar 6. PMID 17367656
- [Background] Chakravarty T, Henry TD, Kittleson M, Lima J, Siegel RJ, Slipczuk L, Pogoda JM, Smith RR, Malliaras K, Marban L, Ascheim DD, Marban E, Makkar RR. Allogeneic cardiosphere-derived cells for the treatment of heart failure with reduced ejection fraction: the Dilated cardiomYopathy iNtervention with Allogeneic MyocardIally-regenerative Cells (DYNAMIC) trial. EuroIntervention. 2020 Jul 17;16(4):e293-e300. doi: 10.4244/EIJ-D-19-00035. PMID 31763984
- [Background] Tseliou E, Kanazawa H, Dawkins J, Gallet R, Kreke M, Smith R, Middleton R, Valle J, Marban L, Kar S, Makkar R, Marban E. Widespread Myocardial Delivery of Heart-Derived Stem Cells by Nonocclusive Triple-Vessel Intracoronary Infusion in Porcine Ischemic Cardiomyopathy: Superior Attenuation of Adverse Remodeling Documented by Magnetic Resonance Imaging and Histology. PLoS One. 2016 Jan 19;11(1):e0144523. doi: 10.1371/journal.pone.0144523. eCollection 2016. PMID 26784932